CLINICAL TRIAL: NCT04321070
Title: A Randomized, Double-Blind, Multiple Center Placebo Controlled Study Comparing Taro Product to RLD and Both Treatments to a Placebo Control in the Treatment of Acne Vulgaris
Brief Title: Bio-equivalence Study With Clinical Endpoints in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLPL 1907
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Clindamycin Phosphate (Experimental): Topical, once daily, for 84 days.
  Interventions: Drug: Clindamycin Phosphate
- Clindamycin Phosphate RLD (Active Comparator): Topical, once daily, for 84 days
  Interventions: Drug: Clindamycin Phosphate RLD
- Vehicle of the test product (Placebo Comparator): Topical, once daily, for 84 days
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Clindamycin Phosphate — A thin film of investigation product will be applied to the affected areas of the face once daily
  Other Names: Lotion
  Arms: Clindamycin Phosphate
Drug: Clindamycin Phosphate RLD — A thin film of investigation product will be applied to the affected areas of the face once daily
  Other Names: Lotion
  Arms: Clindamycin Phosphate RLD
Drug: Placebos — A thin film of investigation product will be applied to the affected areas of the face once daily
  Other Names: Vehicle
  Arms: Vehicle of the test product

SUMMARY:
Bio-equivalence Study With Clinical Endpoints in the Treatment of Acne Vulgaris

DETAILED DESCRIPTION:
Randomized, Double-Blind, Multiple Center Placebo Controlled Study Comparing Taro Product to RLD and Both Treatments to a Placebo Control in the Treatment of Acne Vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non pregnant female aged ≥ 12 and ≤ 40years with a clinical diagnosis of acne vulgaris.
* Subjects who are 18 years of age or older (up to the age of 40) must have provided IRB approved written informed consent.
* Subjects must have a definite clinical diagnosis of acne vulgaris severity grade 2, 3, or 4 as per the Investigator's Global Assessment (IGA).

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning to become pregnant during study participation
* Subjects with a history of hypersensitivity or allergy to adapalene, retinoids and/or any of the study medication ingredients, have a known hypersensitivity to adapalene and benzoyl peroxide and its excitements.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 550 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Demonstration of Bioequivalence | Week 12
  Demonstration of Bioequivalence in percent change in inflammatory and non-inflammatory lesion counts

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Yantovskiy, Study Director — Taro Pharmaceuticals, Inc.
Locations (1):
- Catawba Research LLC, Charlotte, North Carolina, United States